CLINICAL TRIAL: NCT04176016
Title: Safety Study of Radiolabeled (111In or 90Y) OTSA101-DTPA, an Anti-Frizzled Homolog 10 (FZD10) Monoclonal Antibody, to Evaluate Safety and Pharmacokinetics in Patients With Relapsed or Refractory Synovial Sarcoma
Brief Title: Phase I Study of Radiolabeled OTSA101-DTPA in Patients With Relapsed or Refractory Synovial Sarcoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Some of the raw materials for the investigational drug are difficult to obtain and expensive.
Sponsor: OncoTherapy Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTS3050102
Record Dates: First submitted 2019-11-20; First posted 2019-11-25 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Relapsed or Refractory Synovial Sarcoma
MeSH Terms: conditions — Recurrence; Sarcoma, Synovial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Study Arm, no competitor (Experimental)
  Interventions: Drug: OTSA101-DTPA-111In; Drug: OTSA101-DTPA-90Y

INTERVENTIONS:
Drug: OTSA101-DTPA-111In — single IV injection, 185MBq/body
Drug: OTSA101-DTPA-90Y — IV injection (max. 3 injections per patient), 1110MBq/body

SUMMARY:
The purpose of this study is to evaluate safety and pharmacokinetics as well as the biodistribution of OTSA101-DTPA-111In and to evaluate the safety of intravenous administration of OTSA101-DTPA-90Y.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a documented relapsed or refractory synovial sarcoma after standard chemotherapy
2. Patients ≥18 years of age at the time of obtaining informed consent
3. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
4. Patients with measurable lesion
5. Patients not received any anti-malignancy agent or specified surgical intervention within 28 days or specified radiotherapy within 14 days prior to study registration.
6. Patients without any clinically significant laboratory abnormality.
7. Patients with adequate heart function as measured by echocardiography or multiple gated acquisition scan (MUGA).
8. Patients with adequate pulmonary function as measured by pulmonary function tests.
9. Patients who are either not of childbearing potential or who agree to use a contraception method during the study and for 12 months after the last dose of study drug
10. Patients must be able to understand and be willing to sign a written informed consent

Exclusion Criteria:

1. Patients with documented concurrent malignancy.
2. Patients with brain metastasis with clinical symptoms.
3. Patients with any infection requiring systemic treatment.
4. Patients with lung inflammation or pulmonary fibrosis.
5. Patients with a known history of hypersensitivities to antibody agents or serum albumin agents.
6. Patients with a known history of autoimmune diseases.
7. Patients with myocardial infarction (MI) within 6 months prior to study registration.
8. Patients with uncontrolled diseases.
9. Patients with any disease requiring continuous systemic administration of steroids or immunosuppressants.
10. Patients with evidence of active HBV, HCV or HIV infection.
11. Pregnant or breastfeeding female patients, or female patients with suspected pregnancy.
12. Patients who are participating any other investigational treatments during the study.
13. Patients with psychiatric disorders and is considered to have difficulty to study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) and Biodistribution of OTSA101-DTPA-111In | up to 72 hours post dosing
  Concentration of OTSA101-DTPA in plasma and the distribution of OTSA101-DTPA in the body by imaging scan will be assessed.
Safety of OTSA101-DTPA-111In | up to 10 days post dosing
  This outcome will be evaluated via overall listing of Treatment-Emergent Adverse Events and the incidence of each Treatment-Emergent Adverse Event that meets DLT criteria.
Safety of OTSA101-DTPA-90Y | up to 6 weeks post dosing
  This outcome will be evaluated via overall listing of Treatment-Emergent Adverse Events and the incidence of each Treatment-Emergent Adverse Event that meets DLT criteria.

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Osaka International Cancer Institute, Osaka
  - Cancer Institute Hospital of JFCR, Tokyo
  - National Cancer Center Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No